CLINICAL TRIAL: NCT05187546
Title: An Open Label, Single Center Study to Evaluate the Safety and Test-retest Characteristics of [18F]PI-2620 as PET Radioligand for Imaging Tau Deposition in the Brains of Patients With Progressive Supranuclear Palsy Richardson Syndrome (PSP-RS) Compared to Non-demented Controls (NDC)
Brief Title: Test-retest Study With [18F]PI-2620 in PSP-RS and NDC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Life Molecular Imaging GmbH (Industry)
Responsible Party: Sponsor
Organization: Life Molecular Imaging SA (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: LMT-02-01-21
Record Dates: First submitted 2021-11-23; First posted 2022-01-12 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Progressive Supranuclear Palsy
Keywords: Tau PET; [18F]PI-2620; Test-retest; Progressive Supranuclear Palsy
MeSH Terms: conditions — Supranuclear Palsy, Progressive | interventions — ((18)F)PI-2620

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Imaging characteristics of [18F]PI-2620 for detection of Tau deposition in the brain of PSP patients (Experimental): All eligible PSP patients will receive two injections of the investigational imaging agent [18F]PI-2620: at a baseline PET imaging session and at a follow-up PET imaging session to evaluate the test-retest imaging characteristics. 10 PSP patients will be required to complete the study arm.
  Interventions: Drug: [18F]-PI2620
- Imaging characteristics of [18F]PI-2620 for detection of Tau deposition in the brain of NDC subjects (Experimental): All eligible non-demented control (NDC) subjects will receive two injections of the investigational imaging agent [18F]PI-2620: at a baseline PET imaging session and at a follow-up PET imaging session to evaluate the test-retest imaging characteristics. 5 NDC subjects will be required to complete the study arm.
  Interventions: Drug: [18F]-PI2620

INTERVENTIONS:
Drug: [18F]-PI2620 — [18F]PI-2620 is a radioactive diagnostic agent being developed for the indication of PET imaging of the brain to detect tau pathology in adult patients who are being evaluated for neurodegenerative decline. All patients will receive two administrations of [18F]PI-2620 at a radioactive dose of 185 megabecquerel (MBq).

SUMMARY:
The overall goal of this protocol is to evaluate the imaging characteristics of [18F]PI-2620 using positron emission tomography (PET) in patients with progressive supranuclear palsy, Richardson's syndrome (PSP-RS)

DETAILED DESCRIPTION:
The imaging characteristics of [18F]PI-2620 using positron emission tomography (PET) in patients with progressive supranuclear palsy, Richardson's syndrome (PSP-RS) will be evaluated by a) determining the test-retest variability of the [18F]PI-2620 binding parameters in brain of patients with PSP-RS and non-demented controls (NDC).

ELIGIBILITY:
Inclusion Criteria (for all subjects)

* Males and females aged 50-80 years
* Able to understand, sign and date written informed consent
* Signed and dated written informed consent obtained from the subject
* The subject has an appropriate caregiver capable of accompanying subject, if necessary
* Have an Montreal Cognitive Assessment (MoCa) score ≥ 27
* Female subjects must be documented by medical records or physician's note to be either surgically sterile (by means of hysterectomy, bilateral salpingectomy or bilateral oophorectomy) or post-menopausal for at least 1 year (no menses for 12 months without an alternative medical cause). If they are of child-bearing potential, must commit to use of a highly effective contraceptive measure for the duration of the study
* Male subjects and their partners of childbearing potential must commit to the use of a highly effective method of contraception for a minimum of 90 days following each PET scan
* Male subjects must commit to not donate sperm for a minimum of 90 days after each PET scan
* Willing and able to cooperate with study procedures including lying flat and still on the scanning bed for 60 minutes

Inclusion criteria for non-demented controls (NDC)

* Healthy with no clinically relevant finding on physical examination at screening
* No cognitive impairment from neuropsychological battery as judged by the investigator
* A brain MRI without evidence of significant neurological pathology
* A beta-amyloid Neuraceq® PET demonstrating a negative beta-amyloid status
* No signs of movement disorder as judged by Progressive Supranuclear Palsy Rating Scale (PSPRS), Movement Disorder Society - Unified Parkinson's Disability Rating Scale (MDS-UPDRS) and Progressive Supranuclear Palsy Clinical Deficits Scale (PSP-CDS)

Inclusion Criteria for patients with probable PSP-RS

* Patients with a clinical diagnosis of probable PSP-RS based on the Movement Disorder Society criteria (Höglinger et al., 2017)
* Medications taken for symptomatic treatment of PSP must be maintained on a stable dosage regimen for at least 30 days before the [18F]PI-2620 PET imaging visits

Exclusion Criteria (for all subjects)

* Hemoglobin value < 10 g/dL
* Laboratory tests with clinically significant abnormalities and/or clinically significant unstable medical illness equivalent to CTC v5.0 (common toxicity criteria) toxicities greater than grade 2
* Evidence of clinically significant disease that is expected to interfere with cognitive assessments or the ability to complete the study procedures
* Subjects with clinically significant renal and hepatic dysfunction as judged by the investigator
* Known hypersensitivity to the active substance or to any of the excipients of [18F]PI-2620
* Known hypersensitivity to the active substance or to any of the excipients of Neuraceq®, for NDC only
* Subject has received an investigational drug including treatments targeting Amyloid-beta or tau within 3 months of screening
* Pregnant (or having the intention of getting pregnant), lactating or breastfeeding
* Unsuitable veins for repeated venipuncture.
* Subject has a contraindication to blood sampling and/or arterial cannulation, including but not limited to peripheral vascular disease, Raynaud's phenomenon as determined by abnormal Allen's test or abnormal coagulation profile at screening
* MRI exclusion criteria include but not limited to: Findings of cerebrovascular disease (more than two lacunar infarcts, any territorial infarct >1 cm3, or deep white matter abnormality corresponding to an overall Fazekas scale of 3 with at least one confluent hyperintense lesion on the Fluid-Attenuated Inversion Recovery (FLAIR) sequence that is 20 mm in any dimension), infectious disease, space-occupying lesions, normal pressure hydrocephalus or any other abnormalities associated with Central Nervous System (CNS) disease
* Implants such as implanted cardiac pacemakers or defibrillators, insulin pumps, cochlear implants, metallic ocular foreign body, implanted neural stimulators, CNS aneurysm clips and other medical implants that have not been certified for MRI, or history of claustrophobia in MRI
* Unwilling and/or unable to cooperate with study procedures

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-03-05 (Actual)

PRIMARY OUTCOMES:
Test-retest variability of the [18F]PI-2620 binding parameters in brain of patients with PSP-RS and non-demented controls | The duration of the study for participants may be up to 74 days
  Test-retest variability of [18F]PI-2620 accumulation will be analyzed using quantification
Number of adverse events | The duration of the study for participants may be up to 74 days
  Safety will be evaluated by collection of Adverse Events.

SECONDARY OUTCOMES:
Compare quantification in terms if test-retest variability in PSP-RS and NDC | The duration of the study for participants may be up to 74 days
  Comparison of quantification in terms of test-retest variability in PSP and NDC. The ability of [18F]PI-2620 to discriminate between PSP-RS and NDC will be assessed.
Correlate radioligand binding in PSP-RS with clinical scales | The duration of the study for participants may be up to 74 days
  Correlation of radioligand binding with clinical scales in PSP-RS will be analyzed

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Stephens, MD, PhD, Study Director — Life Molecular Imaging; Matthias Brendel, MD, Principal Investigator — Department of Nuclear Medicine, University of Munich
Locations (1):
- Ludwig-Maximilians-Universität München, Munich, Germany

IPD SHARING:
Plan to Share IPD: No